CLINICAL TRIAL: NCT01342289
Title: Shortened-duration Tacrolimus Following Nonmyeloablative, Related Donor BMT With High-dose Posttransplantation Cyclophosphamide
Brief Title: Shorter Course Tacrolimus After Nonmyeloablative, Related Donor BMT With High-dose Posttransplantation Cyclophosphamide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J1151; NA_00048378 (Other: JHMIRB)
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Hodgkin's Lymphoma; Leukemia; Myelodysplastic Syndrome(MDS); Multiple Myeloma; Non Hodgkin's Lymphoma
Keywords: Nonmyeloablative; Allogeneic; Bone Marrow Transplant (BMT); Tacrolimus; Cyclophosphamide
MeSH Terms: conditions — Hodgkin Disease; Leukemia; Myelodysplastic Syndromes; Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Whole-Body Irradiation; Mycophenolic Acid; Tacrolimus; Bone Marrow Transplantation

STUDY DESIGN:
Intervention Model Description: Participants were initially enrolled on the 90-day arm. When that arm completed enrollment, participants were enrolled on the 120-day arm while safety of the 90-day arm was evaluated. The 90-day arm was found to be safe, so participants were then enrolled on the 60-day arm for the remainder of the study.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tacrolimus 60 (Experimental): Non-myeloablative bone marrow transplant with fludarabine, cyclophosphamide, total body irradiation conditioning regimen and cyclophosphamide, mycophenolate mofetil, and tacrolimus prophylaxis for graft-versus-host disease (GVHD). Tacrolimus was given for 60 days.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total body irradiation; Drug: Mycophenolate Mofetil; Drug: Tacrolimus 60; Biological: Bone marrow transplant
- Tacrolimus 90 (Experimental): Non-myeloablative bone marrow transplant with fludarabine, cyclophosphamide, total body irradiation conditioning regimen and cyclophosphamide, mycophenolate mofetil, and tacrolimus prophylaxis for graft-versus-host disease (GVHD). Tacrolimus was given for 90 days.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total body irradiation; Drug: Mycophenolate Mofetil; Drug: Tacrolimus 90; Biological: Bone marrow transplant
- Tacrolimus 120 (Experimental): Non-myeloablative bone marrow transplant with fludarabine, cyclophosphamide, total body irradiation conditioning regimen and cyclophosphamide, mycophenolate mofetil, and tacrolimus prophylaxis for graft-versus-host disease (GVHD). Tacrolimus was given for 120 days.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total body irradiation; Drug: Mycophenolate Mofetil; Drug: Tacrolimus 120; Biological: Bone marrow transplant

INTERVENTIONS:
Drug: Cyclophosphamide — Days -6 and -5: 14.5 mg/kg/day IV. Days 3 and 4: 50 mg/kg/day IV.
  Other Names: Cytoxan
Drug: Fludarabine — Days -6, -5, -4, -3, and -2: 30 mg/m^2/day IV.
  Other Names: Fludara
Radiation: Total body irradiation — Day -1: 200 centigray in one fraction.
  Other Names: TBI
Drug: Mycophenolate Mofetil — Days 5 to 35: 15 mg/kg PO three times per day; max daily dose 1 g.
  Other Names: MMF; CellCept
Drug: Tacrolimus 60 — Begin dosing at 1 mg IV daily on Day 5. Dose is titrated according to serum levels. Stop at Day 60.
  Other Names: FK-506; Prograf
  Arms: Tacrolimus 60
Drug: Tacrolimus 90 — Begin dosing at 1 mg IV daily on Day 5. Dose is titrated according to serum levels. Stop at Day 90.
  Other Names: FK-506; Prograf
  Arms: Tacrolimus 90
Drug: Tacrolimus 120 — Begin dosing at 1 mg IV daily on Day 5. Dose is titrated according to serum levels. Stop at Day 120.
  Other Names: FK-506; Prograf
  Arms: Tacrolimus 120
Biological: Bone marrow transplant — Donor stem cells infused IV on Day 0.
  Other Names: BMT

SUMMARY:
This research is being done to learn more about nonmyeloablative bone marrow transplantation (BMT), also known as a "mini" transplant for patients with blood cancers, using bone marrow from a relative.

DETAILED DESCRIPTION:
The main goal is to learn whether a drug called tacrolimus, which is an immune-lowering drug (an immunosuppressant) given after transplant to help prevent certain complications, can be given safely for a shorter period of time than it has been in the past.

At the present time there are few or no cures for your type of disease outside of a bone marrow transplant. The bone marrow for this transplant comes from a relative who is a half-match or "haplo" match to you. Possible donors include parents, siblings, and children. In order to help the bone marrow grow, or "take", inside your body, you will receive chemotherapy and radiation before the transplant. After the transplant you will receive high doses of cyclophosphamide (Cytoxan®) along with other medications to lower the immune system, tacrolimus. These medications may lower the risk of graft versus host disease (GVHD) and of your body rejecting the bone marrow graft.

ELIGIBILITY:
Inclusion Criteria:

1. 0.5-75 years
2. Suitable first-degree related, HLA haploidentical or HLA-matched donor
3. Eligible diagnoses:

   a. Low-grade non-Hodgkin's lymphoma or plasma cell neoplasm with either of the following, and with stable disease or better prior to transplantation: i. Progressed during multiagent therapy, failed at least two prior therapies (excluding single agent rituximab), or there is evidence of prior transformation ii. SLL or CLL with 11q or 17p deletion or with progression < 6 months after a purine analog-containing regimen

   b. Relapsed, refractory, or progressive aggressive non Hodgkin's lymphoma (including mantle cell lymphoma), with PR or better prior to transplantation, and autologous BMT is not recommended. Note: Patients with Burkitt's, atypical Burkitt's, or acute lymphoblastic lymphoma must be in CR.

   c. Relapsed, refractory, or progressive Hodgkin's lymphoma meeting one of the following criteria, and autologous BMT is not recommend: i. PR or better prior to transplantation. ii. Stable disease prior to transplantation, provided that the disease is low-volume and disease control is regarded as sufficient to proceed with BMT. Eligibility of such patients will be determined on a case-by-case basis with the PI or co-PI.

   d. One of the following poor-risk lymphomas or plasma cell neoplasms, in PR or better prior to transplantation: i. Transformed lymphoma ii. T-cell PLL iii. Peripheral T-cell lymphoma iv. NK or NK/T-cell lymphoma v. Blastic/blastoid mantle cell lymphoma vi. Plasma cell leukemia

   e. For patients with SLL, CLL, or PLL, < 20% of bone marrow cellularity involved by this process (to lower risk of graft rejection).

   f. Relapsed, refractory, or progressive acute leukemia in second or subsequent remission, with remission defined as <5% bone marrow blasts morphologically.

   g. Poor-risk acute leukemia in first remission, with remission defined as <5% bone marrow blasts morphologically: i. AML with at least one of the following: AML arising from MDS or a myeloproliferative disorder, or secondary AML Presence of Flt3 internal tandem duplications Poor-risk cytogenetics Primary refractory disease ii. ALL (leukemia and/or lymphoma) with at least one of the following: Poor-risk cytogenetics Clear evidence of hypodiploidy Primary refractory disease iii. Biphenotypic leukemia

   h. MDS with at least one of the following poor-risk features: i. Poor-risk cytogenetics ii. IPSS score of INT-2 or greater iii. Treatment-related or secondary MDS iv. MDS diagnosed before age 21 years v. Progression on or lack of response to standard DNA-methyltransferase inhibitor therapy vi. Life-threatening cytopenias, including those requiring frequent transfusions

   i. Interferon- or imatinib-refractory CML in first chronic phase, or CML in second or subsequent chronic phase

   j. Philadelphia chromosome negative myeloproliferative disease (including myelofibrosis)

   k. Chronic myelomonocytic leukemia

   l. Juvenile myelomonocytic leukemia
4. One of the following:

   1. Cytotoxic chemotherapy, alemtuzumab, or an adequate course of 5-azacitidine or decitabine must have been given within 3 months prior to start of conditioning or
   2. Previous BMT within 6 months prior to start of conditioning. --Note: Patients who have received treatment outside of these windows may be eligible if it is deemed sufficient to reduce graft rejection risk; this will be decided on a case-by-case basis by the PI or co-PI.

Exclusion Criteria:

1. Active extramedullary leukemia or known active Central Nervous System (CNS) involvement by malignancy.
2. Previous Bone marrow transplant (BMT) less than 3 months prior to start of conditioning.
3. Inadequate end-organ function as measured by:

   1. Left ventricular ejection fraction less than or equal to 35% or shortening fraction less than 25%
   2. Bilirubin greater than or equal to 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and ALT and AST greater than or equal to 5 x ULN
   3. FEV1 and FVC less than or equal to 40% of predicted; or if unable to perform pulmonary function tests due to young age, oxygen saturation less than 92% on room air
4. Previous allogeneic BMT (syngeneic BMT permissible).
5. Pregnant or breast-feeding.
6. Uncontrolled infection.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety of reduced-dose tacrolimus as assessed by Percentage of Participants with severe graft versus host disease (GVHD) | Day 5 - Day 120
  Percentage of participants with severe graft versus host disease (GVHD) defined as grade III-IV acute GVHD or extensive chronic GVHD. Acute GVHD is defined by the Przepiorka criteria, which stages the degree of organ involvement in the skin, liver, and gastrointestinal (GI) tract, based on severity, with Stage 1+ being least severe and stage 4+ being the most severe. Grading of acute GVHD is as follows: Grade I (skin involvement stages 1+ to 2+, with no liver or GI involvement), Grade II (skin involvement stages 1+ to 3+, liver 1+, GI tract 1+), Grade III (skin involvement stages 2+ to 3+, liver 1+, GI tract 2+ to 4+), Grade IV (skin involvement stages 4+, Liver 4+). Chronic GVHD is defined by the NIH consensus criteria. This system gives scores from 0 to 3 for Karnofsky performance score, skin, mouth, eyes, gastrointestinal, liver, lungs, joints, and genitals, as well as an overall severity. Higher scores indicate more severe disease. Scores are not totaled or added up.
Tolerability of tacrolimus as assessed by percentage of participants with treatment-emergent adverse events | Up to 120 days
  Percentage of participants with grade 3-4 toxicity by CTCAE 4.0 attributable to tacrolimus.

SECONDARY OUTCOMES:
Percentage of participants experiencing acute GVHD | Up to 7 years
  Percentage of participants with grade II-IV and III-IV acute GVHD. Acute GVHD is defined by the Przepiorka criteria, which stages the degree of organ involvement in the skin, liver, and gastrointestinal (GI) tract, based on severity, with Stage 1+ being least severe and stage 4+ being the most severe. Grading of acute GVHD is as follows: Grade I (skin involvement stages 1+ to 2+, with no liver or GI involvement), Grade II (skin involvement stages 1+ to 3+, liver 1+, GI tract 1+), Grade III (skin involvement stages 2+ to 3+, liver 1+, GI tract 2+ to 4+), Grade IV (skin involvement stages 4+, Liver 4+).
Percentage of participants experiencing chronic GVHD | Up to 7 years
  Percentage of participants with chronic GVHD. Chronic GVHD is defined by the NIH consensus criteria. This system gives scores from 0 to 3 for Karnofsky performance score, skin, mouth, eyes, gastrointestinal, liver, lungs, joints, and genitals, as well as an overall severity (mild, moderate, or severe). Higher scores indicate more severe disease. Scores are not totalled or added up.
Disease relapse | Up to 7 years
  Percentage of participants experiencing disease relapse or progression.
Non-relapse mortality | Up to 7 years
  Percentage of participants who died for any reason other than disease relapse or progression.
Use of immunosuppression | Up to 2 years
  Percentage of participants who: required use of steroids; required use of non-steroid immunosuppression; and who were able to discontinue immunosuppression after starting treatment.
Survival | Up to 7 years
  Percentage of participants who are alive with and without disease relapse or progression.
Chimerism | 30 and 60 days
  Percentage of participants who had >=95% donor chimerism.
Engraftment | 30 and 60 days
  Percentage of participants who had successful engraftment of neutrophils and platelets.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jones, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kasamon YL, Fuchs EJ, Zahurak M, Rosner GL, Symons HJ, Gladstone DE, Huff CA, Swinnen LJ, Brodsky RA, Matsui WH, Borrello I, Shanbhag S, Cooke KR, Ambinder RF, Luznik L, Bolanos-Meade J, Jones RJ. Shortened-Duration Tacrolimus after Nonmyeloablative, HLA-Haploidentical Bone Marrow Transplantation. Biol Blood Marrow Transplant. 2018 May;24(5):1022-1028. doi: 10.1016/j.bbmt.2018.01.011. Epub 2018 Jan 17. PMID 29353109

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-05-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT01342289/Prot_SAP_000.pdf